CLINICAL TRIAL: NCT01562990
Title: A Multi-center, Phase IB/II, Open Label, Single Arm Study of Inotuzumab Ozogamicin Plus Rituximab (R-CMC544) Alternating With Gemcitabine-oxaliplatin Plus Rituximab(R-GEMOX)in Patients Aged From 18 to 80 Years With CD20 and CD22 Positive Diffuse Large B-cell Lymphoma (DLBCL) in Relapse After/Refractory to 1ST or 2ND Line Treatment, Who Are no Candidates for Autologous Transplant.
Brief Title: Phase Ib/II Study of the Efficacy and Safety of the R-CMC544/R-GEMOX Combination in Diffuse Lage B-cell Lymphoma at First or Second Relapse
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Lymphoma Academic Research Organisation (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMC-R-GEMOX; 2011-003849-18 (EudraCT Number)
Record Dates: First submitted 2012-03-20; First posted 2012-03-26 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-05

CONDITIONS: Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Inotuzumab Ozogamicin; Gemcitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- R-CMC544 and R-GEMOX (Experimental): Treatment with R-CMC544 and R-GEMOX
  Interventions: Drug: Rituximab, CMC544, Gemcitabine and Oxaliplatine

INTERVENTIONS:
Drug: Rituximab, CMC544, Gemcitabine and Oxaliplatine — 2 cycles of induction of 56 days each, starting with the administration of R-CMC544 on day 1, followed by the administration of R-GEMOX on day 29 and 43.
  2 cycles of consolidation of 56 days each, starting with the administration of R-CMC544 on day 1, followed by the administration of R-GEMOX on day 29 and 43.

SUMMARY:
The purpose of this study is to determine the recommended dose of CMC544 administered in combination with rituximab (R-CMC544), and in alternance with rituximab, gemcitabine and oxaliplatin (R-GEMOX) in the first phase of the study. After that, efficacy and safety of this combination will be evaluated preliminarily in patients with DLBCL in relapse or refractory, who are no candidates for autologous transplant.

DETAILED DESCRIPTION:
This study is a multicenter, phase Ib/II, open-label, single arm trial evaluating the efficacy and safety of R-CMC544 alternated with R-GEMOX in patients with CD20 and CD22 positive DLBCL in relapse after/refractory to 1st or 2nd line treatment, who are no candidates for autologous transplant.

The study consists of 2 phases. In part 1 (potential dose de-escalation phase) subjects will be enrolled at a fixed dose of CMC544. In case of occurrence of dose limiting toxicity (DLT), cohorts of 3 to 6 subjects will evaluate a de-escalating dose of CMC544 in combination with set doses of rituximab, gemcitabine and oxaliplatin in order to obtain the MTD or recommended dose of CMC544 in this regimen. In part 2 (dose expansion phase) further safety and preliminary efficacy data of the proposed combination will be analyzed.

All patients will receive two 56 day induction cycles of alternating R-CMC544 (given on day 1) and R-GEMOX (given on day 29 and 43). Patients who obtain CR or PR, will then go on a consolidation of another two 56 day cycles of alternating R-CMC544 (given on day 1) and R-GEMOX (given on day 29 and 43).

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented CD20 and CD22 positive diffuse large B-cell lymphoma, according to WHO classification. CD20 and CD22 immunophenotyping at initial diagnosis is acceptable. If such prior documentation is not available, then the immunophenotyping at relapse must be established by fine-needle aspirate or biopsy or by circulating CD20 and CD22 positive NHL cells from peripheral blood during screening. Upon registration the pathological report confirming the diagnosis, must be available
* In first or second relapse or refractory to first and/or second line treatment. Refractory is defined as having exhibited less than or PR to a prior rituximab containing regimen or having relapsed within 6 months of the last dose of a prior rituximab containing regimen.
* Measurable disease by bidimensional transverse CT scan assessment
* Not eligible for autologous transplantation.
* Previously treated with a chemotherapy regimen containing anthracyclines and rituximab.
* Aged 18 - 80 years.
* ECOG performance status 0 to 2.
* Minimum life expectancy of 3 months.
* Signed written informed consent.

Exclusion Criteria:

* Burkitt, mantle cell and T-cell lymphomas.
* Central nervous system or meningeal involvement by the lymphoma.
* Contraindication to any drug contained in the R-GEMOX combination chemotherapy.
* Treatment with any investigational drug within 30 days before the first planned cycle of chemotherapy and during the study.
* Nitrosurea or mitomycin C administration within 6 weeks prior to study start.
* Major debulking surgery within 3 weeks of treatment.
* Any of the following lab abnormalities (unless related to the lymphoma or bone marrow infiltration):

Absolute neutrophil count (ANC) < 1.500/µL (1,5.109/L).

Platelet count < 100.000/µL (100.109/L).

Creatinin level > 150 µmol/L (1,7 mg/dL) or 1,5 - 2,0x ULN.

Total bilirubin level > 30 µmol/L (1,8 mg/dL) or 1,5x ULN.

Serum AST/SGOT or ALT/SGPT >2,5x ULN.

* Documented infection with HIV, active hepatitis B or C infection.
* Any serious active disease or co-morbid medical condition that, according to the investigator's decision, will substantially increase the risk associated with the subject's participation in the study. Prior history of malignancies other than lymphoma with the exception of non-melanoma skin tumors (basal cell or squamous cell carcinoma of the skin) or stage 0 (in situ) cervical carcinoma unless the subject has been disease-free for 5 or more years..
* LVEF less than 50% (measured by echocardiography or scintigraphy).
* Previous myocardial infarction or pulmonary hypertension within 6 months before the first dose of investigational product.
* Congestive heart failure NYHA stage III or IV
* Known chronic liver disease (eg. Cirrhosis) or suspected alcohol abuse.
* Pregnant or lactating females
* Men and women who are biologically capable of having children not willing to use an adequate method of birth control during the study and up to 18 months after the last dose of investigational product.
* Adult patient unable to provide informed consent because of intellectual impairment, any serious medical condition, laboratory abnormality or psychiatric illness.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-12; Primary Completion 2014-08 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Determination of the Recommended Dose of R-CMC544 | Up to 16 weeks
  Determination of recommended dose will be based on safety parameters and particularly on incidence of DLTs

SECONDARY OUTCOMES:
OVERALL RESPONSE RATE | Up to 32 weeks
  Assessment of response will be based on the International Workshop to Standardize Response criteria for NHL (Criteria for evaluation of response in Non-Hodgkin's lymphoma (Cheson, 1999 and 2007). Patient is defined as a responder if he/she has a complete response (CR) or partial response (PR) at the end of treatment. A descriptive analysis will also be performed considering as non-responders all patients who relapsed or died during treatment phase even if they were prematurely withdrawn as responder
PROGRESSION-FREE SURVIVAL | Up to 3.5 years
  Progression-Free Survival will be measured from the date of inclusion to the date of first documented disease progression, relapse or death from any cause. Responding patients and patients who are lost to follow up will be censored at their last tumor assessment date.
EVENT FREE SURVIVAL | Up to 3.5 years
  Event-Free Survival will be measured from the date of inclusion to the date of first documented disease progression, relapse, initiation of new anti-lymphoma therapy or death from any cause. Responding patients and patients who are lost to follow up will be censored at their last tumor assessment date.
OVERALL SURVIVAL | Up to 3.5 years
  Overall survival will be measured from the date of inclusion to the date of death from any cause. Patients who are alive at the time of analysis will be censored at the date of the last contact.
COMPLETE RESPONSE RATE | 30 or 32 weeks (depending on induction cycle length)
  Assessment of response will be based on the International Workshop to Standardize Response criteria for NHL (Criteria for evaluation of response in Non-Hodgkin's lymphoma (Cheson, 2007)).
  Patient without response assessment (due to whatever reason) will be considered as nonresponder.

CONTACTS AND LOCATIONS:
Overall Officials: Fritz OFFNER, MD, Study Chair — Lymphoma Study Association; Corinne HAIOUN, PhD, Study Chair — Lymphoma Study Association
Locations (11):
- Belgium (3):
  - AZ Sint Jan, Bruges
  - University Hospital Gent, Ghent
  - CHU Mont-Godinne, Yvoir
- France (8):
  - Hôpital Henri Mondor, Créteil
  - CHU de Dijon, Dijon
  - CHRU de Lille, Lille
  - CHU Lyon - Sud, Lyon
  - CHU Hôtel Dieu, Nantes
  - CHU Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
  - CHU Brabois, Vandœuvre-lès-Nancy

REFERENCES:
- See also: LYSA (Lymphoma Study Association) website — http://lysa-lymphoma.com/